CLINICAL TRIAL: NCT05227001
Title: A PHASE 1, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLIND, DOSE-FINDING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF SELF-AMPLIFYING RNA VACCINE PREPARATIONS AGAINST INFLUENZA IN HEALTHY INDIVIDUALS
Brief Title: A Study To Learn About The Study Vaccine (Called Self-Amplifying Ribonucleic Acid (RNA)) For The Prevention of Influenza
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4861001
Record Dates: First submitted 2022-01-19; First posted 2022-02-07 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Influenza, Human
Keywords: Grippe; Flu; Influenza; Vaccine; RNA vaccine; Self-amplifying
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (26):
- PF-07852352 Influenza saRNA, low dose (Experimental)
  Interventions: Biological: PF-07852352 Influenza saRNA 1
- PF-07852352 Influenza saRNA, mid dose (Experimental)
  Interventions: Biological: PF-07852352 Influenza saRNA 1
- PF-07852352 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07852352 Influenza saRNA 1
- PF-07836391 Influenza saRNA, low dose (Experimental)
  Interventions: Biological: PF-07836391 Influenza saRNA
- PF-07836391 Influenza saRNA, mid dose (Experimental)
  Interventions: Biological: PF-07836391 Influenza saRNA
- PF-07836391 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07836391 Influenza saRNA
- PF-07836394 Influenza saRNA, low dose (Experimental)
  Interventions: Biological: PF-07836394 Influenza saRNA
- PF-07836394 Influenza saRNA, mid dose (Experimental)
  Interventions: Biological: PF-07836394 Influenza saRNA
- PF-07836394 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07836394 Influenza saRNA
- PF-07836395 Influenza saRNA, low dose (Experimental)
  Interventions: Biological: PF-07836395 Influenza saRNA
- PF-07836395 Influenza saRNA, mid dose (Experimental)
  Interventions: Biological: PF-07836395 Influenza saRNA
- PF-07836395 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07836395 Influenza saRNA
- PF-07836396 Influenza saRNA, low dose (Experimental)
  Interventions: Biological: PF-07836396 Influenza saRNA
- PF-07836396 Influenza saRNA, mid dose (Experimental)
  Interventions: Biological: PF-07836396 Influenza saRNA
- PF-07836396 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07836396 Influenza saRNA
- PF-07867246 Influenza saRNA, mid dose (Experimental)
  Interventions: Biological: PF-07867246 Influenza saRNA
- PF-07867246 Influenza saRNA, low dose (Experimental)
  Interventions: Biological: PF-07867246 Influenza saRNA
- PF-07867246 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07867246 Influenza saRNA
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Quadrivalent influenza vaccine (QIV) (Active Comparator)
  Interventions: Biological: Quadrivalent influenza vaccine (QIV)
- PF-07871987 Influenza saRNA, low dose (Experimental)
  Interventions: Biological: PF-07871987 Influenza saRNA
- PF-07871987 Influenza saRNA, mid dose (Experimental)
  Interventions: Biological: PF-07871987 Influenza saRNA
- PF-07871987 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07871987 Influenza saRNA
- PF-07914705 Influenza saRNA mid dose (Experimental)
  Interventions: Biological: PF-07914705 Influenza saRNA
- PF-07914705 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07914705 Influenza saRNA
- PF-07915048 Influenza saRNA, high dose (Experimental)
  Interventions: Biological: PF-07915048 Influenza saRNA

INTERVENTIONS:
Biological: PF-07852352 Influenza saRNA 1 — Intramuscular injection
  Arms: PF-07852352 Influenza saRNA, high dose; PF-07852352 Influenza saRNA, low dose; PF-07852352 Influenza saRNA, mid dose
Biological: PF-07836391 Influenza saRNA — Intramuscular injection
  Arms: PF-07836391 Influenza saRNA, high dose; PF-07836391 Influenza saRNA, low dose; PF-07836391 Influenza saRNA, mid dose
Biological: PF-07836394 Influenza saRNA — Intramuscular injection
  Arms: PF-07836394 Influenza saRNA, high dose; PF-07836394 Influenza saRNA, low dose; PF-07836394 Influenza saRNA, mid dose
Biological: PF-07836395 Influenza saRNA — Intramuscular injection
  Arms: PF-07836395 Influenza saRNA, high dose; PF-07836395 Influenza saRNA, low dose; PF-07836395 Influenza saRNA, mid dose
Biological: PF-07836396 Influenza saRNA — Intramuscular injection
  Arms: PF-07836396 Influenza saRNA, high dose; PF-07836396 Influenza saRNA, low dose; PF-07836396 Influenza saRNA, mid dose
Biological: PF-07867246 Influenza saRNA — Intramuscular injection
  Arms: PF-07867246 Influenza saRNA, high dose; PF-07867246 Influenza saRNA, low dose; PF-07867246 Influenza saRNA, mid dose
Biological: Placebo — Intramuscular injection
  Arms: Placebo
Biological: Quadrivalent influenza vaccine (QIV) — Intramuscular injection
  Arms: Quadrivalent influenza vaccine (QIV)
Biological: PF-07871987 Influenza saRNA — Intramuscular injection
  Arms: PF-07871987 Influenza saRNA, high dose; PF-07871987 Influenza saRNA, low dose; PF-07871987 Influenza saRNA, mid dose
Biological: PF-07914705 Influenza saRNA — Intramuscular injection
  Arms: PF-07914705 Influenza saRNA mid dose; PF-07914705 Influenza saRNA, high dose
Biological: PF-07915048 Influenza saRNA — Intramuscular injection
  Arms: PF-07915048 Influenza saRNA, high dose

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study vaccine for the potential prevention of influenza. The study vaccine is called Self-Amplifying Ribonucleic Acid vaccine (saRNA vaccine). This study is seeking participants who:

* Are between the age of 18 to 49 years old.
* Are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Are healthy as determined by medical history, physical examinations, and the study doctor.
* For male participants, can father children and willing to use an acceptable method of contraception. Female participants who are not of childbearing potential; or male participant not able to father children.
* Are capable of giving signed informed consent. Participants will receive either the saRNA vaccine, a licensed Influenza Vaccine (QIV) or a placebo. Participants will not know which vaccine they receive in advance. A placebo does not have any medicine in it but looks just like the study medicine. Participants will receive the study vaccines as a single shot in the arm. We will compare participant experiences to help us determine if the saRNA vaccine is safe and effective. Participants will take part in this study for 6 months. During this time, they will receive the study vaccine and participate in follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 to 49 years of age.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Male participant who is able to father children and willing to use an acceptable method of contraception; or female participant not of childbearing potential; or male participant not able to father children.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Allergy to egg proteins (egg or egg products) or chicken proteins.
* Participant who has had significant exposure to laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 infection), coronavirus disease 2019 (COVID-19), or influenza in the past 14 days known prior to Visit 1
* Any participant who has a SARS-CoV-2 RT-PCR or antigen test in the past 10 days prior to Visit 1 that has not been confirmed as negative.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or planned receipt throughout the study.
* Vaccination with any influenza vaccine within 6 months (175 days) before study intervention administration.
* Any participant who has received or plans to receive a nucleoside-modified messenger ribonucleic acid (modRNA)-platform SARS-CoV-2 vaccine within 60 days of Visit 1
* Previous vaccination with an saRNA or an alphavirus replicon vaccine preparation.
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
* Screening hematology/blood chemistry lab >=Grade 1 abnormality. Except Bilirubin, other stable Grade1 abnormalities may be considered eligible by Investigator.
* Screening electrocardiogram (ECG) that is consistent with probable or possible myocarditis or pericarditis, or demonstrates clinically relevant abnormalities that may affect participant safety or study results.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Participation in strenuous or endurance exercise through Visit 3.
* Prior history of heart disease.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 442 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting local reactions | For 10 days after vaccination
  Pain at the injection site, redness, and swelling, as self-reported in electronic diaries.
Percentage of participants reporting systemic events | For 10 days after vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain, as self reported in electronic diaries.
Percentage of participants reporting adverse events | From vaccination to 4 weeks after vaccination
  As elicited by investigational site staff.
Percentage of participants reporting serious adverse events | From vaccination to 6 months after vaccination
  As elicited by investigational site staff.
Percentage of participants with abnormal hematology and chemistry laboratory values | 2 days after vaccination
  As measured at the central laboratory
Percentage of participants with abnormal hematology and chemistry laboratory values | 1 week after vaccination
  As measured at the central laboratory
Percentage of participants with grading shifts in hematology and chemistry laboratory assessments | Between baseline and 2 days after vaccination
  As measured at the central laboratory.
Percentage of participants with grading shifts in hematology and chemistry laboratory assessments | Between baseline and 1 week after vaccination
  As measured at the central laboratory
Percentage of participants with new electrocardiogram (ECG) abnormalities | 2 days after vaccination
  ECG abnormalities consistent with probable or possible myocarditis or pericarditis, as judged by a cardiologist
Percentage of participants with new ECG abnormalities | 1 week after vaccination
  ECG abnormalities consistent with probable or possible myocarditis or pericarditis, as judged by a cardiologist

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) of hemagglutination inhibition (HAI) titers | At Baseline, and 1-, 2- and 4-weeks after vaccination
  As measured at the central laboratory
Geometric mean fold rise (GMFR) in HAI titers from before vaccination to each subsequent timepoint | At Baseline, and 1-, 2- and 4-weeks after vaccination
  As measured at the central laboratory
Proportion of participants achieving HAI seroconversion for each strain | At 1-, 2-, and 4-weeks after vaccination
  As measured at the central laboratory
Proportion of participants with HAI titer >=1:40 for each strain | At Baseline, and 1-, 2-, and 4-weeks after vaccination
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (25):
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Finlay Medical Research, Greenacres City, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Mount Sinai Hospital, Miami Beach, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - Pinnacle Health Care Center, Pembroke Pines, Florida
  - Comprehensive Cardiology Consultants, Pembroke Pines, Florida
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Pioneer Heart Institute, Lincoln, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - SUNY Upstate Medical University Global Health Laboratory, Syracuse, New York
  - SUNY Upstate Medical University Institute for Global Health, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Benchmark Research, Austin, Texas
  - Eric S. Tiblier, MD, Austin, Texas
  - DM Clinical Research, Tomball, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4861001